CLINICAL TRIAL: NCT03437382
Title: HOlmium Radioembolization as Adjuvant Treatment to Radiofrequency Ablation for Early STage Hepatocellular Carcinoma (HORA EST HCC)
Brief Title: Holmium Radioembolization as Adjuvant Treatment to RFA for Early Stage HCC: Dose Finding Study
Acronym: HORA EST HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Health Holland (Other); Quirem Medical B.V. (Industry); Medtronic (Industry); Maag Lever Darm Stichting (Other)
Responsible Party: Principal Investigator, MCBurgmans, Principle Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P17.161; ZonMW (Other Grant/Funding Number: PTO 2017 - 40-41200-98-9286)
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: HCC; Early Stage HCC
Keywords: Hepatocellular carcinoma; Radiofrequency ablation (RFA); Radioembolization; Quirem Spheres; Selective internal radiation therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: single-arm, interventional, dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RFA + radioembolization (Other): Quirem Medical Holmium-166 radioembolization microspheres
  Interventions: Device: Quirem Medical Holmium-166 radioembolization microspheres

INTERVENTIONS:
Device: Quirem Medical Holmium-166 radioembolization microspheres — radioembolisation as adjuvant treatment to RFA

SUMMARY:
In this multi-center, dose-finding study, patients with early stage hepatocellular carcinoma according to the Barcelona Clinic Liver Cancer (BCLC) staging system will be included to receive percutaneous radiofrequency ablation in combination with RFA with adjuvant segmental radioembolization.

DETAILED DESCRIPTION:
RFA + adjuvant radioembolsation with Quirem Spheres

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age > 18 years
* Single HCC lesion with diameter of ≥ 2-5cm or up to three lesions with each lesion measuring no more than 3cm (confined to one lobe)
* HCC diagnosis is based on histology or non-invasive imaging criteria according to EORTC-EASL guidelines
* Child Pugh A or B ≤7
* ECOG performance status ≤ 2
* Bilirubin < 2mg/dL
* ASAT < 5x upper limit of normal
* ALAT < 5x upper limit of normal
* Thrombocytes ≥ 50 X 10^9/L

Exclusion Criteria:

* Recurrent HCC
* Tumor location precluding percutaneous RFA
* Bilobar tumor involvement
* Vascular tumor invasion or extrahepatic metastasis
* Hemihepatectomy
* Severe comorbidity (e.g. cardiovascular disease, diabetes with nephropathy, active infections)
* Uncorrectable coagulopathy
* Large arterio-portovenous shunt
* Previous radiotherapy to the liver
* Surgical hepatico-enterostomy
* Hepatic resection with placement of surgical clips that may cause artefacts on MRI
* Incompetent/ mentally disabled
* Pregnancy, inadequate anticonception
* Calculated lung dose >30Gy
* Creatinine clearance < 50 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Dose-finding | 1 year
  Treatment area dose that will result in delivery of a radiation absorbed dose of ≥ 120Gy to the target area in at least 90% of patients.

SECONDARY OUTCOMES:
Toxicity | 1 year
  Toxicity of RFA with adjuvant segmental radioembolization as assessed by complications according to CTCAE v4.0
Local tumor recurrence | 6 months and 12 months
  Local tumor recurrence at 6 months as assessed by multiphase CT or dynamic MRI
Time to progression | 1 year
  time until disease progresses
Progression-free survival | 1 year
  Kaplan-Meier analysis of progression free survival
Quality of Life | Throughout the first year after treatment.
  Quality of Life will be assessed by means of the EORTC QLQ HCC-18 questionnaire
Quality of Life | Throughout the first year after treatment.
  Quality of Life will be assessed by means of the C-30 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hendriks P, Rietbergen DDD, van Erkel AR, Coenraad MJ, Arntz MJ, Bennink RJ, Braat AE, Crobach S, van Delden OM, Dibbets-Schneider P, van der Hulle T, Klumpen HJ, van der Meer RW, Nijsen JFW, van Rijswijk CSP, Roosen J, Ruijter BN, Smit F, Stam MK, Takkenberg RB, Tushuizen ME, van Velden FHP, de Geus-Oei LF, Burgmans MC; Dutch Hepatocellular and Cholangiocarcinoma Group. Adjuvant holmium-166 radioembolization after radiofrequency ablation in early-stage hepatocellular carcinoma patients: a dose-finding study (HORA EST HCC trial). Eur J Nucl Med Mol Imaging. 2024 Jun;51(7):2085-2097. doi: 10.1007/s00259-024-06630-z. Epub 2024 Feb 8. PMID 38329507
- [Derived] Hendriks P, Rietbergen DDD, van Erkel AR, Coenraad MJ, Arntz MJ, Bennink RJ, Braat AE, Crobach ASLP, van Delden OM, van der Hulle T, Klumpen HJ, van der Meer RW, Nijsen JFW, van Rijswijk CSP, Roosen J, Ruijter BN, Smit F, Stam MK, Takkenberg RB, Tushuizen ME, van Velden FHP, de Geus-Oei LF, Burgmans MC; Dutch Hepatocellular Cholangiocarcinoma Group. Study Protocol: Adjuvant Holmium-166 Radioembolization After Radiofrequency Ablation in Early-Stage Hepatocellular Carcinoma Patients-A Dose-Finding Study (HORA EST HCC Trial). Cardiovasc Intervent Radiol. 2022 Aug;45(8):1057-1063. doi: 10.1007/s00270-022-03162-7. Epub 2022 May 26. PMID 35618860